CLINICAL TRIAL: NCT03774563
Title: Sleep During Weight Loss and Weight Loss Maintenance
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jessica.K.Salwen-Deremer, Clinical Psychologist, Phd, Dartmouth-Hitchcock Medical Center
Other Study IDs: D19005
Record Dates: First submitted 2018-11-16; First posted 2018-12-13 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Sleep; Weight Loss
Keywords: weight loss; sleep
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to examine the changes of sleep during weight loss and weight loss management. The research staff will also obtain data on sleep disturbances, insomnia symptoms, risk of sleep apnea, circadian preferences, weight loss self-efficacy, emotional eating, executive functioning, loneliness and social isolation, and patients' beliefs about how sleep might impact their weight control or vice versa.

DETAILED DESCRIPTION:
This study is an observational study using a longitudinal data collection design with non-invasive measures. Fifty participants who are about to begin the Healthy Lifestyle Program (HLP) at the Weight and Wellness Clinic (WWC) and another 50 participants who are about to complete HLP will be recruited to the study. After informed consent is obtained, the patient will be asked to complete several questionnaires about sleep and wellbeing. Their height and weight will also be measured by the research staff. The patient will then be given a wrist-worn accelerometer to wear for 16 weeks to measure their sleep and physical activity. They will be asked to complete the same set of questions at approximately the 8th and 16th week at a research visit. Data on existing diagnosis of sleep disorders will be extracted from the patients' electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Adult overweight or obese patients who are enrolled in or who completed the Healthy Lifestyle Program at Weight and Wellness Center.Exclusion Criteria:

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals who are about to begin the Healthy Lifestyle Program at the Weight and Wellness Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Change in sleep duration | Week 1 and 16th week
  Sleep parameters measured by the ActiGraph model wGT3X-BT, a wrist-accelerometer. Measured in minutes of sleep per night. Higher number indicating longer sleep duration. Change from week 1 to week 16 will be measured.
Changes in physical activity | Week 1 and 16th week
  Measured by the Actigraph model wGT3X-BT, a wrist accelerometer. Measured in minutes of moderate to vigorous activity.
Change in sleep quality | Week 1, 8th week, and 16th week
  Pittsburgh Sleep Quality Index (PSQI) will be used to assess a range of sleep disturbances including insomnia, sleep-related breathing difficulties, and use of sleep aids. A total score of 5 or more is indicative of poor sleep quality. Possible score range is 0-21.
Change in Severity of Insomnia | Week 1, 8th week, and 16th week
  Insomnia Severity Index (ISI) will be used to assess the severity of insomnia symptoms and subjective daytime impairments.The total score ranges from 0 to 63, with higher scores indicating more severe anxiety symptoms.
Change in Risk for sleep apnea | Week 1, 8th week, and 16th week
  The STOP-BANG Questionnaire will be used to assess the patient's risk for sleep apnea. Scores range from 0-8. The higher the score indicates an increase in the probability of sleep apnea.
Change in Peak alertness | Week 1, 8th week, and 16th week
  The Morningness-Eveningness Questionnaire (MEQ) will be used to assess whether the patient's circadian rhythm produces peak alertness in the morning or the evening. Multiple choice, 4-5 point scale. The sum gives a score ranging from 16 to 86; scores of 41 and below indicate "evening types", scores of 59 and above indicate "morning types", scores between 42-58 indicate "intermediate types".
Change in self-efficacy in one's ability to lose or maintain weight | Week 1, 8th week, and 16th week
  The Weight Loss Self-Efficacy Scale will be used to assess self-efficacy in one's ability to lose or maintain weight. Measured by subjective rating percentages of confidence, 0-100%. The higher the percentage the higher the ability to maintain or lose weight.
Change in strategies to lose weight | Week 1, 8th week, and 16th week
  The Weight Control Strategies Scale will be used to assess strategies used to lose weight. The sum of scores ranges from 0-120. The higher the scores the more strategies being used to lose weight.
Change in emotional and disinhibited eating | Week 1, 8th week, and 16th week
  Three Factors Eating Questionnaire will be used to measure emotional and disinhibited eating. Comprised of 18 items , which are aggregated to three separate scale scores. A 4-point response format is used.
Mood symptoms | Week 1, 8th week, and 16th week
  will be assessed using the Patient Healthy Questionnaire (PHQ9). The PHQ9 scores range from 0-27, with lower numbers indicating minimal to no depression and higher numbers indicating severe depression.
Change in Delayed Discounting Index | Week 1, 8th week, and 16th week
  Executive functioning will be assessed using the delay discounting task and the response disinhibition task. K index corresponding to the degree to which a participant discounts future rewards compared to immediate rewards. Will be computed based on a validated algorithm.
Change in social isolation | Week 1, 8th week, and 16th week
  Social isolation will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) isolation scale. The PROMIS scale has six items each with a response options ranging in value from one to five. The lowest possible score is 6 and highest possible score is 30.
Anxiety symptoms | Week 1, 8th week, and 16th week
  will be assessed using the Generalized Anxiety Disorder-7 (GAD7). The GAD7 scores range from 5-21, with 5-9 indicating mild, 10-14 moderate, and greater than 15 severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Wai S Chan, Phd, Principal Investigator — Dartmouth College; Sivan Rotenberg, Phd, Principal Investigator — Dartmouth College; Jessica K Salwen-Deremer, Phd, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

DOCUMENTS (1):
  • Study Protocol (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT03774563/Prot_000.pdf